CLINICAL TRIAL: NCT06862934
Title: Liver Transplantation for Unresectable Intrahepatic Colangiocarcinoma After Sustained Response to Neoadjuvant Treatments (iCOLA)
Brief Title: Liver Transplantation for Unresectable Intrahepatic Colangiocarcinoma After Sustained Response to Neoadjuvant Treatments
Acronym: iCOLA
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 253-24
Record Dates: First submitted 2025-01-27; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-01

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc)
Keywords: liver transplantation; transarterial radioembolization; downstaging
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and transplant specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Transplant: Patients enrolled within the study who undergo downstaging and liver transplantation after with various combinations of chemotherapy +/- immunotherapy and TARE
- Controls 1 (unresectable): Historical controls with the same inclusion criteria as the iCOLA protocol, treated with systemic and locoregional therapies and prospectively recruited patients with tumor response who refused transplantation or were not found eligible to LT for medical/non-oncological conditions
- Controls 2 (resectable): Patients with resectable iCC who underwent curative-intent liver resection, matched to the transplanted patients using demographic characteristics, tumor burden and pre-surgical therapies

SUMMARY:
This is single-arm, observational, academic, investigator-driven study investigating the efficacy of liver transplantation after successful and sustained downstaging/tumor control of liver-limited unresectable intrahepatic cholangiocarcinoma. The downstaging protocol includes chemotherapy +/- immunotherapy and transarterial radioembolization (TARE) with Yttrium-90 in various combinations.

DETAILED DESCRIPTION:
This is a single-arm, observational, academic, investigator-driven study investigating the efficacy of liver transplantation after successful and sustained downstaging/tumor control of liver-limited unresectable intrahepatic cholangiocarcinoma.

Patients with biopsy-proven unresectable ICC who fit within inclusion criteria will be enrolled in the study. Patients with unresectable ICC who enter the protocol with an intention-to-treat strategy will first undergo CT scan +/- MRI, FDG-PET and staging laparoscopy with nodal sampling at the hepatic hilum (at least stations 8 and 12). In case of negative staging (no peritoneal carcinomatosis, no tumor spread in lymph nodes, negative tumor citology in the peritoneal washing), they will receive downstaging with state-of-the-art chemotherapy +/- immune checkpoint inhibitors (ICIs) (at the time of writing: gemcitabine-cisplatin +/- durvalumab) for 2 cycles, followed by transarterial radioembolization with Y90 (Y90-TARE), followed by at least 4 other cycles of gemcitabine-cisplatin +/- durvalumab. If actionable mutations are present at gene sequencing of tumoral tissue are present, molecular-targeted treatments with FGFR-inhibitors, IDH-1 inhibitors and PARP-inhibitors are allowed after multidisciplinary evaluations. Patients who cannot undergo Y90-TARE due to absolute contraindications (e.g., evidence of pulmonary shunts at angioscintigraphy) may be considered for stereotactic body radiation therapy (SBRT).

After downstaging, patients will undergo disease restaging with CT scan +/- MRI, FDG-PET and CA19-9 and, if at least tumor stability is confirmed with CA19-9 < 200 u/ml, they will undergo transplant screening and listing.

Both naive patients and patients already receiving systemic and/or locoregional therapies for their unresectable ICC are eligible as long as sustained response is demonstrated. In all instances, they will undergo staging laparoscopy and, if negative (see above) with at least 6 months of tumor stability from diagnosis, they will go directly to transplant screening and listing.

During listing, restaging will be performed every two months with CT scan and/or MRI, molecular markers and FDG-PET. Maintenance therapy is allowed at the discretion of the patient's oncology team. The target interval between listing and transplant should be less than 90 days.

Tumor response will be determined according to RECIST, mRECIST and Choi criteria.

In case of disease progression during listing, the patient will be suspended from the transplant waiting list. Re-listing is allowed after second-line therapy if disease stability for at least four months if achieved, at the discretion of the multidisciplinary tumor and transplant board of INT Milan.

Any kind of donor will be considered as suitable for the recruited patients, including marginal marginal organ donation (DCD, split-liver, age >75, severe steatosis, etcetera).

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of iCCA (biopsy-proven tumor)
* Either first diagnosis or post-resection recurrence (occurring ≥ 6 months after resection)
* Unresectability assessment due to tumor location (leading to insufficient live remnant with/out implementation of hypertrophic parenchymal techniques) or underlying liver disease. Non-resectability assessed by an expert surgical team with experience on both resection and transplantation (centralized at INT Milan).
* Age between 18 and 70 years
* No macrovascular tumor invasion (NB: portal vein and/or hepatic vein occlusion from the external tumor compression and classified as "encasement" could be considered after expert radiology review)
* No extrahepatic spread
* Disease stability for at least 6 months
* CA 19-9 < 200 u/ml at transplant listing in absence of jaundice
* No medical and surgical contraindications to liver transplantation
* Good performance status, Eastern Cooperative Oncology Group (ECOG) 0 or 1
* No concomitant malignancies or history of other malignancies in the previous 5 years
* Written informed consent

Exclusion Criteria:

* Hilar and distal cholangiocarcinoma
* Progression of disease under chemotherapy +/- radiation therapy, assessed with either RECIST, mRECIST or Choi criteria
* Evidence of lymph-nodal metastases
* Evidence of extrahepatic disease
* Prior extrahepatic metastatic disease
* Concomitant malignancies or history of other malignancies in the previous 5 years
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any reason why, in the opinion of the investigator, the patient should not participate to the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable liver-limited intrahepatic cholangiocarcinoma with no non-oncological contraindications to liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival vs unresectable patients | 3 years
  OS at 3 years after liver transplant will be matched and compared with OS of patients with similar characteristics that were not offered LT, taken from an institutional historical series and from patients found not eligible to LT due to medical/non-oncological conditions

SECONDARY OUTCOMES:
3-year recurrence-free survival vs unresectable patients | 3 years
  To evaluate the time to recurrence after LT in patients with unresectable iCCA, RFS at 3 years after LT will be matched and compared with time to progression of patients with similar characteristics that were not offered LT, taken from an institutional historical series and from patients found non-eligible to LT due to medical/non-oncological conditions
90-day morbidity | 90 days and long-term
  The safety of chemotherapy +/- immunotherapy, locoregional treatments and liver transplatation in patients with unresectable iCCA will be assessed with the Clavien-Dindo classification and the Comprehensive Complication Index
Quality of life | 3 years
  The impact of this treatment strategy and of LT on quality of life in patients with unresectable iCCA will be assessed with validated questionnaires. Questionnaires will be performed at baseline and at 6 months intervals; they will be matched and compared with that of eligible patients recruited within the same study period and receiving non-transplant treatments.
3-year OS vs resectable patients | 3 years
  OS after LT in patients with unresectable iCCA will be compared with OS of patients with similar characteristics, but with resectable tumors, who underwent surgical resection during the same time period
3-year DFS vs resectable patients | 3 years
  DFS after LT in patients with unresectable iCCA will be compared with DFS of patients with similar characteristics, but with resectable tumors, who underwent surgical resection during the same time period

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori di Milano, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maspero M, Sposito C, Bongini MA, Cascella T, Flores M, Maccauro M, Chiesa C, Niger M, Pietrantonio F, Leoncini G, Bellia V, Bhoori S, Mazzaferro V. Liver Transplantation for Intrahepatic Cholangiocarcinoma After Chemotherapy and Radioembolization: An Intention-To-Treat Study. Transpl Int. 2024 Oct 31;37:13641. doi: 10.3389/ti.2024.13641. eCollection 2024. PMID 39544321